CLINICAL TRIAL: NCT01846377
Title: Video Games for Obesity and Diabetes Prevention: Efficacy Trial
Brief Title: Video Games for Obesity and Diabetes Prevention-Diab & Nano
Acronym: G4H-DiabNano
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Thomas Baranowski, Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-29172
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: video game; diet; physical activity; sedentary behavior; obesity; diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Motor Activity; Sedentary Behavior; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G4H-Diab-Nano (Experimental): Intervention - play two videogames Diab and Nanoswarm (9 sessions each, 18 total sessions) over a 12-week time period.
  Interventions: Behavioral: G4H-Diab-Nano
- Wait List Control (No Intervention): 5-months after baseline assessment they will receive the two video games: 1) Diab and 2) Nanoswarm.

INTERVENTIONS:
Behavioral: G4H-Diab-Nano — The Diab and Nanoswarm games present fun, challenging: knowledge mini-games enabling children to learn desired behavior changes; goal-setting tailored to child's current behaviors and preferences to make lifestyle changes; problem solving to enable children to find strategies to overcome behavior change barriers; motivational statements tailored to child's values to enhance their desire to make the goal related lifestyle changes; and energy balance games to enable them to balance food portions with physical activities. Each game has 9 sessions each with approximately 45-60 min of game-play. At the end of each session, goals are set. The child is allowed to re-play non-behavior change mini-games, and view video segments, but not redo their goal setting or behavior change mini-games.
  Arms: G4H-Diab-Nano

SUMMARY:
With the increasing rates of child obesity and diabetes, innovative programs are needed that capture children's attention and permit behavior change messages to get through. Serious video games with their immersive stories offer one such promising alternative due to their low cost approach to intervention since the games have already been developed, and can be broadly disseminated by simply reproducing and distributing their DVDs. While using video games for health promotion is controversial, this study will establish whether video games can effectively change diabetes and obesity risks (especially fasting insulin, diet and physical activity) among children.

"Escape from Diab" and "Nanoswarm: Invasion from Inner Space" are two video games that targeted children to increase fruit, vegetable and water intakes, reduce sedentary behaviors (SB), and increase physical activity in a pilot study with a relatively low risk children. In light of this, it is important to test whether these games can help decrease diabetes (i.e. fasting insulin) and obesity risks with high risk (85%tile < BMI < 99%tile) 10 to 12 year old children.

Children will be randomly assigned to treatment or control groups. The treatment group will play "Diab" and "Nano" over a 3-month time period. A wait-list control group will receive the "Diab" and "Nano" games at the end of their second post assessment (5-months post baseline assessment).

DETAILED DESCRIPTION:
This project is to conduct an efficacy trial of Diab and Nanoswarm to assess their potential for minimizing T2D and obesity risks. The proposed research will be conducted in two phases, covering a 3-year period: implementation and evaluation phase of 2.5 years and an analysis phase of 0.5 years.

Specific Aim 1: Conduct an efficacy outcome evaluation of Diab and Nano using a randomized clinical trial.

Hypothesis 1: Children will decrease fasting insulin by, at least, 2μU/dl, increase FV intake by at least 1.0 servings/day, and increase MVPA by at least 10 min/day from baseline to up to 3 months post baseline.

Hypothesis 2: Diet, MVPA and fasting insulin changes will not be moderated by demographic characteristics (e.g. gender, age, ethnic group).

Hypothesis 3: Fasting insulin change will be mediated by changes in diet, PA and SB.

Hypothesis 4: Diet and PA change outcomes will be mediated by changes in child's preferences and intrinsic motivation for FV and PA.

Control Intervention will be a wait list group and receive the intervention at the end of the 5-month post assessment.

Intervention: Children will play the games at home. Each game session should take about 45 to 60 minutes to complete with an ability to go back and replay the non-behavior mini-games.

Child Measures include:

* Fasting insulin and glucose
* Height, weight and waist circumference
* Body mass index (BMI; kg/m2) BMI %
* Fruit, vegetable and beverage intake by food frequency, and preferences, self efficacy, and intrinsic motivation
* Physical activity (PA) by Actigraph GT3X accelerometer and PA preferences/enjoyment, self efficacy, intrinsic motivation and home equipment availability
* Transportation/immersion/liking of video games played
* Social desirability to reflect giving answers that are socially acceptable or expected

Parent Measures includes:

* Family demographics
* Food and physical activity equipment availability at home
* Report of if their child liked and played the video games

ELIGIBILITY:
Inclusion criteria:

* Children who are 10-12 years of age
* with a 85th%tile to 99th%tile BMI
* willing to complete all measures including providing a blood sample and
* having internet access and a computer with these minimum requirements:
* Operating System: Microsoft Windows XP (SP3), Windows Vista (SP2), Windows 7 (SP1), Windows 8 or 8.1 Processor: 2.13 GHz Intel Core 2 Duo E6400 or 2.8 GHz AMD Athlon 64 x2 5600+ minimum System Memory: 2Gbytes RAM Screen Resolution: 1280 x 800 minimum Hard Drive: 10Gbytes minimum free space Sound: Sound card with speakers or headphone jack DVD Optical Drive (needed for installation only) DirectX Runtimes: (October 2006 version or newer) Internet: Broadband Connection Computer Manufactured after 2009.

Exclusion Criteria:

* Child does not speak English (since both games are in English),
* has a medical condition that influences diet, physical activity, obesity, or the ability to complete questionnaires,
* has type 2 diabetes mellitus;
* does not have a qualified computer and internet access at home.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in fasting insulin from baseline to immediate post intervention (approximately 3 months post baseline assessment) and 2-months post intervention (approximately 5 months post baseline assessment) | Three time points: baseline, post intervention (approximately three months post baseline), two month post intervention (approximately 5 months post baseline)

SECONDARY OUTCOMES:
Change in Fruit and Vegetable Intake | Three time points: baseline, post intervention (approximately three months post baseline), two month post intervention (approximately 5 months post baseline)

OTHER OUTCOMES:
Change in Moderate to Vigorous Physical Activity | Three time points: baseline, post intervention (approximately three months post baseline), two month post intervention (approximately 5 months post baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Baranowski, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baranowski T, Baranowski J, Thompson D, Buday R, Jago R, Griffith MJ, Islam N, Nguyen N, Watson KB. Video game play, child diet, and physical activity behavior change a randomized clinical trial. Am J Prev Med. 2011 Jan;40(1):33-8. doi: 10.1016/j.amepre.2010.09.029. PMID 21146765